CLINICAL TRIAL: NCT06421974
Title: A Prospective, Multicenter, Randomized Controlled Trial of the Effectiveness of Robotic Versus Laparoscopic Surgery for Right Colon Cancer
Brief Title: Effectiveness of Robotic Surgery for Right Colon Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang Cancer Hospital (Other); Zhejiang Provincial People's Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Zhangfa Song, Professor, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRRS-ERSRCC
Record Dates: First submitted 2024-05-03; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Colon Cancer; Robotic Surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic surgery for right colon cancer (Experimental): Robot-assisted right colon cancer radical resection group, referred to as robotic surgery group
  Interventions: Procedure: DaVinci si or xi system
- laparoscopic surgery for right colon cancer (Active Comparator): Laparoscopic right colon cancer radical resection group, referred to as laparoscopic surgery group
  Interventions: Procedure: laparoscopic radical resection

INTERVENTIONS:
Procedure: DaVinci si or xi system — In this study, subjects were randomly divided into an experimental group (robot-assisted radical resection of right colon cancer group, referred to as robotic surgery group) and a control group (laparoscopic radical resection of right colon cancer group, referred to as laparoscopic surgery group).
  Arms: Robotic surgery for right colon cancer
Procedure: laparoscopic radical resection — In this study, subjects were randomly divided into an experimental group (robot-assisted radical resection of right colon cancer group, referred to as robotic surgery group) and a control group (laparoscopic radical resection of right colon cancer group, referred to as laparoscopic surgery group).
  Arms: laparoscopic surgery for right colon cancer

SUMMARY:
This study aims to explore through a multi-center, randomized controlled clinical study whether robot-assisted radical resection of right colon cancer is superior to laparoscopic surgery in terms of surgical quality and oncological prognosis.

DETAILED DESCRIPTION:
The incidence rate of colorectal cancer has risen to the second place in my country, highlighting its significant impact on public health. It is a high-incidence malignant tumor that seriously threatens the health of our people. Surgery is the core treatment method for curing colorectal cancer. With the promotion of multidisciplinary comprehensive treatment models, in-depth understanding of abdominal and pelvic anatomy, and innovations in surgical instruments and techniques, colorectal cancer surgery is gradually developing in the direction of minimally invasive and organ function preservation. This advancement not only improves the safety and effectiveness of surgery, but also improves patients' postoperative quality of life. Laparoscopic surgery has obvious minimally invasive advantages in the treatment of right colon cancer. Compared with traditional laparotomy, laparoscopic surgery has the advantages of less trauma, less postoperative pain, faster recovery, and shorter hospital stay.

Since Hohenberger proposed the concept of complete mesocolic excision (CME), the principle of CME has become a key technique in colon cancer surgery, which emphasizes thorough lymph node dissection and precise tumor resection. In radical resection of right colon cancer, CME technology ensures complete resection of surrounding tissue by performing surgery along the natural anatomical plane of blood vessels and nerve plexuses, thereby reducing the local recurrence rate of the tumor. A retrospective cohort study of 1395 cases included in the Danish Colorectal Cancer Study Group showed that the 4-year disease-free survival rate of patients of all stages after CME surgery was 85.8% (95% CI 81.4-90.1), and that after non-CME surgery, the 4-year disease-free survival rate was 85.8% (95% CI 81.4-90.1). The 4-year disease-free survival rate was 75.9% (95% CI 72.2-79.7) (log-rank p=0.0010), which preliminarily proved that the CME principle can significantly improve the disease recurrence-free survival (DFS) rate. This method aims to achieve better tumor cure results through more extensive and complete resection.

However, with the continuous innovation of surgical instruments and technologies, laparoscopic surgery is also facing some challenges. Laparoscopic surgery often provides a two-dimensional field of view, which may limit the surgeon's depth perception and accuracy when performing complex procedures. In addition, the operating rods of traditional laparoscopic tools are relatively long and the operating space is limited, which may lead to difficulties in gesture amplification and fine motor control during surgery, resulting in certain defects in surgical operation accuracy and visual field stability.

The robot-assisted surgical system provides a new technical platform for improving the quality of surgical operations with its enhanced visual capabilities, stable field of view and flexibility of surgical instruments. The stability of the three-dimensional stereo vision system and camera platform can significantly improve the surgical field of view, while the high flexibility of the robotic arm optimizes surgical operations. Existing clinical studies show that compared with traditional laparoscopic surgery, robot-assisted surgical systems have potential advantages in reducing the proportion of conversions to laparotomy, reducing the occurrence of postoperative complications, and shortening postoperative recovery time.

When considering the economic burden of robotic-assisted surgical systems relative to conventional laparoscopic surgery, more rigorous and quantitative evidence is necessary to assess their economic benefits in daily clinical practice. Although robot-assisted surgical systems offer operational advantages, their high equipment investment and maintenance costs remain a major obstacle to their adoption. Therefore, a comprehensive cost-effectiveness analysis, combined with an assessment of surgical outcomes, patient recovery, and long-term health-related quality, is critical to determine its suitability in the healthcare system. The REAL randomized controlled study led by Professor Xu Jianmin compared the surgical quality and long-term tumor prognosis of robot-assisted surgery and conventional laparoscopic surgery in patients with middle and low rectal cancer. The primary endpoint of the study was the 3-year local recurrence rate, while the secondary endpoints focused on the positive circumferential margin rate and the 30-day postoperative complication rate. The short-term secondary endpoint data that have been published so far are encouraging. However, there is still a lack of multicenter randomized controlled clinical studies on the long-term oncological outcomes of robotic surgery for right colon cancer.

This study aims to compare the 3-year disease recurrence-free survival (DFS) between robot-assisted radical right hemicolectomy (RA-LSRHC) and conventional laparoscopic radical right hemicolectomy (LSRHC) through a multicenter, randomized controlled study. The non-inferiority in terms of surgery provides high-quality evidence-based medical evidence for robot-assisted right colon cancer surgery, further optimizes treatment strategies, and improves patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old.
2. ASA classification ≤ Level III.
3. Colon adenocarcinoma was confirmed by colonoscopy and biopsy pathology.
4. Transabdominal enhanced CT showed that the distal and proximal ends of the primary tumor were located in the right colon (cecum to the proximal 1/3 of the transverse colon).
5. Preoperative clinical stage: TanyNanyM0.
6. The patient's condition meets the indications for robotic surgery and is willing to accept the robotic surgery treatment plan.
7. Voluntarily participate in this study and sign the informed consent form. If the subject is unable to read and sign the informed consent form due to incapacity or other reasons, his or her guardian must be responsible for the informed process and sign the informed consent form. If the subject is unable to read the informed consent form (such as illiterate subjects), a witness must witness the informed process and sign the informed consent form.

Exclusion Criteria:

1. Preoperative examination indicates synchronous multiple primary colorectal cancers or other diseases requiring intestinal segmental resection.
2. The results of preoperative imaging examination or intraoperative exploration suggest: 1) The tumor involves surrounding organs and requires combined organ resection; 2) There is distant metastasis; 3) R0 resection cannot be performed.
3. Additional radical surgery after emr and esd surgery.
4. Have a history of any other malignant tumor or familial adenomatous polyposis in the past 5 years, except for cured cervical carcinoma in situ, basal cell carcinoma, papillary thyroid carcinoma or cutaneous squamous cell carcinoma.
5. Combined intestinal obstruction, intestinal perforation, intestinal bleeding, etc. require emergency surgery.
6. Patients who are not suitable for or cannot tolerate robotic or laparoscopic surgery.
7. Pregnant or lactating women.
8. Patients with a history of mental illness.
9. Patients who have received neoadjuvant treatment before surgery.
10. MDT discusses patients who are not suitable for entering the study.
11. Patients who refuse to undergo either robotic or laparoscopic surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The time from randomization to first tumor recurrence/metastasis or death from any cause was defined as the time of last follow-up for patients lost to follow-up(Patients still alive at the end of the study, the end of follow-up).

SECONDARY OUTCOMES:
30-day perioperative complications | up to 1 month.
  Perioperative complications were classified according to the Clavien-Dindo system, including intraoperative, short-term and long-term postoperative complications.
Overall survival | 5-year
  5-year overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shao hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No